CLINICAL TRIAL: NCT04822844
Title: Implementing a Nurse-Driven Aromatherapy Protocol to Decrease the Effect of Postoperative Nausea and Vomiting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: HCA Houston Healthcare Southeast Hospital (Unknown)
Responsible Party: Principal Investigator, Julie George, Director of Surgical Services, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HSC-SN-20-1306
Record Dates: First submitted 2021-03-25; First posted 2021-03-30 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Postoperative Nausea and Vomiting (PONV)
Keywords: aromatherapy
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — lavender oil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aromatherapy with Essential Oil (Experimental): Within 5 minutes of arrival at the PACU, the PACU nurse will proactively offer the patient a 2x2 gauze with two drops of essential oil (patient's choice of ginger or lavender essential oil) for all patients who have opted to participate, regardless of their nausea and vomiting status. Participating patients will continue to use the essential oil during their stay in the PACU, which is typically 45-60 minutes.
  Interventions: Other: Lavender Essential Oil; Other: Ginger Essential Oil

INTERVENTIONS:
Other: Lavender Essential Oil — Within 5 minutes of arrival at the PACU, the PACU nurse will proactively offer the patient a 2x2 gauze with two drops of essential oil (patient's choice of ginger or lavender essential oil) for all patients who have opted to participate, regardless of their nausea and vomiting status. Participating patients will continue to use the essential oil during their stay in the PACU, which is typically 45-60 minutes.
Other: Ginger Essential Oil — Within 5 minutes of arrival at the PACU, the PACU nurse will proactively offer the patient a 2x2 gauze with two drops of essential oil (patient's choice of ginger or lavender essential oil) for all patients who have opted to participate, regardless of their nausea and vomiting status. Participating patients will continue to use the essential oil during their stay in the PACU, which is typically 45-60 minutes.

SUMMARY:
This is a quality improvement project that aims to assess the effect of nurse-driven administration of essential oil aromatherapy on postoperative nausea and vomiting (PONV) in patients while in the post-anesthesia care unit (PACU) after general anesthesia.

DETAILED DESCRIPTION:
In this three-month quality improvement project, nurse-driven aromatherapy will be offered to all patients in the main PACU setting at the Hospital Corporation of America (HCA) Houston Healthcare Southeast Hospital after they have undergone surgical procedures with general anesthesia, with the exception of patients who report allergies or sensitivity to ginger or lavender essential oils (EO) and patients who wish to be excluded from the project.

ELIGIBILITY:
Inclusion Criteria:

* PACU patients who are in the main PACU setting at HCA Houston Healthcare Southeast Hospital after having undergone general anesthesia for a surgical procedure

Exclusion Criteria:

* patients with allergies or sensitivity to ginger or lavender essential oils
* patients who wish to be excluded from the project

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Number of Post-Operative Nausea and Vomiting Episodes While in the PACU | during stay in PACU (about 45-60 minutes)

SECONDARY OUTCOMES:
PACU Length of Stay | time between PACU admission and PACU discharge (about 45-60 minutes)
  PACU length of stay is the time between PACU admission and PACU discharge, measured in minutes.
Number of Participants Who Use Antiemetics While in the PACU | during stay in PACU (about 45-60 minutes)
Patient Satisfaction as Assessed by the Press Ganey Patient Satisfaction Survey | at discharge (about 1 hour after PACU admission)
  The Press Ganey Patient Satisfaction Survey is scored from 0 to 100, with a higher score indicating greater satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Julie George, RN, MSN, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- HCA Houston Healthcare Southeast Hospital, Pasadena, Texas, United States

IPD SHARING:
Plan to Share IPD: No